CLINICAL TRIAL: NCT01870180
Title: Investigating the Efficacy of the MGDRx EyeBag in Patients With Meibomian Gland Dysfunction Related Evaporative Dry Eye
Brief Title: EyeBag Effectiveness in Meibomian Gland Dysfunction
Acronym: MGD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aston University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2013MGD
Record Dates: First submitted 2013-05-24; First posted 2013-06-05 (Estimated); Last update posted 2015-01-15 (Estimated); Status verified 2015-01

CONDITIONS: Meibomian Gland Dysfunction
Keywords: Meibomian Glad Dysfunction; EyeBag; Hot Compress; Dry Eyes
MeSH Terms: conditions — Meibomian Gland Dysfunction; Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- EyeBag (Experimental): Eye self-treated with heated eyebag in the morning and evening each day as per manufacturer's instructions (see http://www.eyebagcompany.com/how)
  Interventions: Device: EyeBag
- Placebo (Placebo Comparator): Non-heated EyeBAG: As with eyebag arm but second eyebag applied on other eye at same time BUT not heated
  Interventions: Other: Placebo

INTERVENTIONS:
Device: EyeBag — fabric bag of beads which can be heated in a microwave
  Other Names: MGDRx EyeBAg
  Arms: EyeBag
Other: Placebo
  Other Names: Non-Heated Eyebag
  Arms: Placebo

SUMMARY:
Meibomian gland dysfunction (MGD) is a common condition that causes the secretion from meibomian glands in the eyelids to become blocked. Normally, the secretion helps to maintain a healthy tear film. In MGD, the tear film becomes unstable and often causes dry eye symptoms. Treatments often involve gently warming the eyelids to melt this blockage which prevents tears from spreading over the eye. Although there has been some research on application of heat with warm moist flannels, the Eye Bags potentially offers a simpler and more effective method of applying heat to the eyelids. This study will test the efficiency of these eyelid warming devices over a period of two weeks use in one eye compared to the other non-treated eye.

DETAILED DESCRIPTION:
Study Design

Contralateral treatment study Randomised eye treated with heated eyebag in the morning and evening each day as per manufacturer's instructions Other eye acts as control with room temperature eyebag overlaid in same manner as treatment eye Investigators masked SMS messaging twice a day for 14 days to remind patients to use eyebag and collect 0-10 comfort score

ELIGIBILITY:
Inclusion Criteria:

* 18 or over
* Have otherwise healthy eyes
* Are prepared not to wear contact lens for the 2 weeks of the trial
* Have a NITBUT <10s
* OSDI score: greater than or equal to 12
* Symptom frequency at least "some of the time"
* Presence of cloudy fluid expressed from at least 1 of the central 8 glands on the lower/upper lid AND/OR presence of poor expressibility from at least 2-3 of the central 8 glands on the lower lid

Exclusion Criteria:

• Blepharitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-05; Primary Completion 2013-07 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in Ocular Symptoms | Between baseline and 2 weeks
  Ocular symptomology: Ocular Surface Disease Index for right and left eyes
Change in Tear Film Quality | Between baseline and 2 weeks
  Non-invasive tear break up time: 3 measurements per eye

SECONDARY OUTCOMES:
Change in Ocular redness | Between baseline and 2 weeks
  Ocular hyperaemia: limbal and temporal conjunctiva for both eyes, images captured
Change in Lipid layer thickness | Between baseline and 2 weeks
  Tear film lipid layer thickness: for right and left eyes, images captured with Tearscope
Change in Meibomian Glands | Between baseline and 2 weeks
  Meibography: for right and left eyes, images captured using Keratograph 5 leading to change in area score

CONTACTS AND LOCATIONS:
Locations (1):
- Aston University, Birmingham, West Midlands, United Kingdom

REFERENCES:
- [Result] Bilkhu PS, Naroo SA, Wolffsohn JS. Randomised masked clinical trial of the MGDRx EyeBag for the treatment of meibomian gland dysfunction-related evaporative dry eye. Br J Ophthalmol. 2014 Dec;98(12):1707-11. doi: 10.1136/bjophthalmol-2014-305220. Epub 2014 Jul 4. PMID 24997178